CLINICAL TRIAL: NCT05023473
Title: Comparison Between Pericapsular Nerve Group Block (Peng) and Morphine Infusion in Reducing the Pain of Proximal Femur Fracture in the Emergency Department, a Randomized Controlled Study
Brief Title: Comparison Between Pericapsular Nerve Group Block (PENG) and Morphine Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PENG block
Record Dates: First submitted 2021-08-14; First posted 2021-08-26 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Analgesia; Femur Fracture
MeSH Terms: conditions — Agnosia; Femoral Fractures | interventions — Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG block+ morhine (Active Comparator): the participants will receive PENG block before being attached to morphine PCA
  Interventions: Procedure: Pericapsular nerve group block; Drug: Morphine Sulfate
- MORPHINE (Active Comparator): The participants will be given morphine PCA without PENG block
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Procedure: Pericapsular nerve group block — patients will receive pericapsular nerve group block
  Arms: PENG block+ morhine
Drug: Morphine Sulfate — morphine will be given to both groups as patient-controlled analgesia PCA

SUMMARY:
The pericapsular nerve group block (PENG) is a regional anaesthetic technique that was developed in 2018, primarily for total hip arthroplasties (THA) as a postoperative analgesia modality with motor sparing benefits.

The block is thought to provide more complete analgesia to the hip by depositing local anaesthetic within the myofascial plane of the psoas muscle and superior pubic ramus.

In this study, the investigators will assess the effect of pericapsular nerve group (PENG) block on pain control in patients with proximal femur fracture in the emergency department.

The Control group will receive morphine as regular patient control analgesia (PCA) The interventional group will receive PENG block before being attached to regular morphine PCA

DETAILED DESCRIPTION:
The pericapsular nerve group block (PENG) is a regional anaesthetic technique that was developed in 2018, primarily for total hip arthroplasties (THA) as a postoperative analgesia modality with motor sparing benefits.

The block is thought to provide more complete analgesia to the hip by depositing local anaesthetic within the myofascial plane of the psoas muscle and superior pubic ramus.

The indications for THA often include degenerative hip disease and traumatic hip fractures. These indications for surgery are relatively common in the elderly population and are associated with significant morbidity and mortality.

Operative intervention, such as THA, has also been associated with significant pain.

Historically, the most commonly performed peripheral nerve blocks include a lumbar plexus block, a femoral nerve block, or a fascia iliaca compartment block to manage post-operative analgesia.

With the understanding that additional articular branches (i.e., from the sciatic nerve) these blocks will provide incomplete analgesia to the hip and may also predispose the patient to fall due to weakness of the quadriceps muscles.

Therefore the ideal block technique should provide complete analgesia of the hip joint and without muscle weakness.

The PENG has been described for postoperative pain control for surgery at the hip joint or the management of post-traumatic pain associated with fractures of the proximal femur/ femoral head.

There are currently no unique contraindications that are specific to the PENG block. Therefore, similar guidelines applicable to most peripheral nerve blocks would apply and include:

* Lack of patient consent
* Skin infection at the site of injection
* Systemic bacteremia or sepsis
* Anticoagulation and antithrombotic medications precautions as detailed by the American society of regional anaesthesia for peripheral nerve blocks The hip joint has a complex innervation, and the pain following hip fractures or total hip arthroplasties is particularly severe. An appropriate plan for perioperative analgesia is challenging, but a multimodal approach including acetaminophen, cox-2 selective NSAIDs, regional anaesthesia, and periarticular infiltration techniques improves patient outcomes.

The ultrasound-guided PENG block allows for coverage of the hip joint, targeting the proximal articular branches that innervate the joint capsule. This proximal approach via ultrasound guidance can confer several advantages over a femoral nerve block by providing more complete analgesia to the hip joint. Additionally, the motor function of the involved extremity should be spared. The PENG block can be used alone as a primary analgesic or in conjunction with other forms of anaesthesia during surgery or in the perioperative period. For lateral surgical incisions, a supplemental lateral femoral cutaneous nerve block provides additional coverage.

With the patient in the supine position, the ultrasound probe is placed on a transverse plane over the anterior superior iliac spine (ASIS). Once the ASIS is identified, the transducer is aligned with the pubic ramus and rotated at approximately 45 degrees, parallel to the inguinal crease. The transducer is then slid medially along this axis until the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), and the psoas tendon is identified, serving as anatomic landmarks.

Sliding the probe distally or gently tilting the caudal will expose the head of the femur. Returning to the initial starting position, a standard 20-22 gauge 100mm needle is inserted in-plane, from lateral to medial, in the plane between the psoas tendon and the pubic ramus. 15-20ml of a long-lasting local anaesthetic ((i.e., 0.5% ropivacaine) is then deposited in this plane, lifting the psoas tendon. Care should be taken to avoid puncturing the psoas tendon. In this study, the investigators will assess the effect of pericapsular nerve group (PENG) block on pain control in patients with proximal femur fracture in the emergency department.

The Control group will receive morphine as regular patient control analgesia (PCA) The interventional group will receive PENG block before being attached to regular morphine PCA

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 18-70 years.
* Patients are ASA I (American Society of Anesthesiology physical status Grade I) = (normal healthy patients) or ASA II (American Society of Anesthesiologists physical status grade II) = (patients with mild systemic disease and no functional limitations).
* Patients having post-traumatic pain associated with fractures of the proximal femur or femoral head.

Exclusion Criteria:

* Patient refusal to participate in the study
* Known allergy to LA.
* Body mass index (BMI) more than 40 kg/m2
* Heart block greater than first degree
* Renal, and hepatic dysfunction
* Underlying coagulopathies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption | immediately at the end of 24 hours
  compare the total morphine consumption in milligrams that is given by patient-controlled analgesia device (PCA)

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | immediately after starting morphine infusion 0,2,4,6,8,10,12,14,16,18,20,22,24 hours at rest
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Incidence of nausea and vomiting | immediately after starting morphine infusion 0,2,4,6,8,10,12,14,16,18,20,22,24 hours at rest
  desire to vomit or actual vomiting as prescribed yeas or no

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided